CLINICAL TRIAL: NCT01998997
Title: A Family Intervention to Decrease Delirium: a Pilot Study
Brief Title: A Family Intervention for Delirium Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monidipa Dasgupta, Associate Professor, Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104385
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Delirium
Keywords: Delirium; Hospitalized elderly
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family educational intervention (Active Comparator): A family educational, non-pharmacologic intervention will be administered to educate family members on how to prevent delirium. Family members will be encouraged to actively participate in this non-pharmacologic intervention.
  Interventions: Behavioral: Family educational intervention
- general health education (Placebo Comparator): The placebo group will be given a brochure on good health habits
  Interventions: Behavioral: Family educational intervention

INTERVENTIONS:
Behavioral: Family educational intervention — The intervention is an educational intervention directed towards delirium prevention specifically for family members of hospitalized seniors. Family members will be encouraged to perform specific interventions that may decrease incident delirium.

SUMMARY:
To address the feasibility of implementing a randomized, educational intervention to prevent delirium, directed at family members of hospitalized older (70 years of age or older) medical in-patients. Specifically rates of recruitment and acceptance rates of such an intervention to family members will be assessed. An estimate of the effect size of this intervention will also be calculated. This is a pilot study. The investigators hypothesize that this intervention will be feasible and agreeable to family members to perform, with acceptance rates exceeding 80%.

DETAILED DESCRIPTION:
In a recent study in Chile, investigators randomized family members of admitted patients to an educational intervention to prevent delirium. Family members actively participated in a non-pharmacological intervention to prevent delirium. This has not been done in a North American environment, with different cultural and climactic factors.

This study will be a randomized controlled trial (pilot study) involving family members. Family members will be randomized to a control group or an educational intervention. The control group will receive a general brochure, outlining general health information published by the Ministry of Health. The intervention group will receive a specific brochure on details around delirium (what it is and how to prevent it), and then a brief educational session comprising a didactic session and to address any questions. This pilot study will examine the feasibility of doing this kind of intervention in a North American environment. The family-based intervention is similar to what was done in the Chilean study. It involves six elements including the educational session. The five other elements include: 1) family being present for extended periods (at least 5 hours if possible); 2) engaging in conversation with study patients for re-orientation to current time and current events; 3) avoiding sensory deprivation (ensuring hearing or visual aids and dentures are available as needed; 4) providing familiar objects to patients; 5) provision of a clock and calendar to the patient. The intervention brochure is similar to what was provided to family members as part of the original Chilean study (kindly provided to the principal investigator, M. Dasgupta, by the lead author of the Chilean study, Dr. F.T. Martinez).

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Residing in the community
* Admitted to a general medical unit at the London Health Sciences center, University Campus
* Having a willing and interested English-speaking family member
* Not delirious on admission
* Able to communicate in English

Exclusion Criteria:

* Terminal condition
* Delirious on admission
* Advanced dementia
* Admission to the ICU (or transfer to the ICU within one week of admission)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
acceptance rate of intervention | 14 weeks
  This is a feasibility study aiming to assess the acceptance of an intervention directed at family members. The acceptance rate will therefore be the primary outcome.

SECONDARY OUTCOMES:
Rate of incident delirium in each of the 2 groups | 14 weeks
  The rate of incident delirium in each of the 2 (control or intervention) groups will be examined in order to calculate the sample size for a future similar intervention study.

OTHER OUTCOMES:
Difficulties in performing the intervention | 14 weeks
  Family members will be surveyed as to what may have been particular difficulties in the intervention to perform. This may help to re-design the intervention for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: monidipa dasgupta, MD, Principal Investigator — Lawson HRI
Locations (1):
- University Hospital, London, Ontario, Canada